CLINICAL TRIAL: NCT01393509
Title: The First-in-human Phase I Trial of PU-H71 in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-041
Record Dates: First submitted 2011-07-09; First posted 2011-07-13 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Solid Tumor; Lymphoma; Myeloproliferative Neoplasms (MPN)
Keywords: PU-H71; Solid Tumor; Lymphoma; 11-041; incurable, locally advanced or metastatic solid tumor malignancy or lymphoma
MeSH Terms: conditions — Neoplasm Metastasis; Lymphoma; Myeloproliferative Disorders | interventions — 9H-purine-9-propanamine, 6-amino-8-((6-iodo-1,3-benzodioxol-5-yl)thio)-N-(1-methylethyl)-

ARMS (1):
- PU-H71 (Experimental): This Phase 1 trial will be an open-label, dose-escalation study of single-agent PU-H71 in patients with advanced solid malignancies and lymphoma.
  Interventions: Drug: PU-H71

INTERVENTIONS:
Drug: PU-H71 — PU-H71 will be administered as an intravenous infusion over 1 hour two times a week on a 2 week on and 1 week off (Q21 day) schedule with a starting dose of 10 mg/m2. A Cycle on study will be defined as 21 days. The same schedule of administration will be used for all patients in this Phase I trial, and a MCRM (modified continual reassessment method)design will be employed. The MPN expansion may explore different dosing schedules.

SUMMARY:
NOTE: This study is now recruiting only patients with Myeloproliferative Neoplasms (MPN). Dose escalation has been completed.

The purpose of this study is to test a new drug, called PU-H71 for the first time in humans, to find out what effects, good or bad, this new drug has on the patient and the cancer at different dose levels. PU-H71 blocks a protein called Heat Shock Protein-90 (Hsp90). Hsp90 is found in both normal and cancer cells, but may be more important in cancer cells. Attacking Hsp90 can stop the function of certain proteins that are needed for cancer cells to survive. The diseases that are part of this study may be especially sensitive to attacking Hsp90, and the investigators have seen signs of disease control in patients with MPN. This study is currently enrolling a cohort expansion for patients with myeloproliferative neoplasms (MPN).

ELIGIBILITY:
Inclusion Criteria:

* The safety-expansion phase will be open to accrual only for patients with MPN.
* ≥ 18 years of age
* For patients with solid malignancies and lymphoma, radiographically detectable (Either FDG-PET, CT scan/ MRI or Bone Scan) or measurable disease will be required. Measurable disease is defined as at least one measurable lesion ≥ 10 mm on CT scan (15 mm for nodal lesions).
* Prior therapy for advanced malignancy with no current curative option
* Neutrophil count ≥ 1,000/μL, platelet count ≥ 50,000/μL, and hemoglobin ≥ 8 g/dL (Platelet count must be assessed at least 7 days after a prior transfusion, if any)
* Serum bilirubin ≤ 1.5 mg/dL;
* AST and ALT≤ 1.5 × ULN
* Serum creatinine ≤ 1.5 mg/dL or creatinine clearance of ≥ 50 mL/min based on a 24-hour urine collection
* Patients receiving hydroxyurea may continue receiving it for up to 14 days after the start of protocol treatment if WBC >30 x10^9/L.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Patients with HIV/AIDS are allowed on study if they have an undetectable viral load, CD4 > 300 and on stable Highly Active Antiretroviral Therapy (HAART) regimen for 1 month.
* Patients who have been treated for at least two weeks with stable doses of corticosteroids to address conditions unrelated to their malignancy will be allowed to continue this treatment during enrollment on the current trial.
* Patients currently being treated with a gonadotropin-releasing hormone agonist (GnRH agonist), bicalutamide or with bisphosphonates may continue treatment while on clinical trial PU-H71 as long as the treatment has been initiated before the study start. GnRH agonist must have been well tolerated for at least three months.
* Optional participation in the microdose imaging trial, IRB#10-139.
* Signed written informed consent and HIPAA consent.
* PATIENTS WITH MPN must be:
* On ruxolitinib for at least three months and on a stable dose for at least 1 month prior to enrollment and taking at least 5 mg twice daily of ruxolitinib
* Tolerating ruxolitinib but with persistent manifestations of disease (i.e. persistent splenomegaly, abnormal blood counts, persistent constitutional symptoms residual fibrosis in bone marrow (2+ or greater), or measurable allele burden as evidenced of clonal JAK2 or MPL mutation).
* Ruxilitinib treatment requirements will be waived for patients who have failed this treatment in the past or for whom this treatment is otherwise contraindicated

EXCLUSION CRITERIA

* Ejection fraction < 50%, as determined by echocardiogram or MUGA scan
* Symptomatic brain or CNS metastases. Previously treated and stable CNS disease is allowed.
* Any of the following for the treatment of cancer within 2 weeks of first study treatment: chemotherapy, immunotherapy, experimental therapy or biologic therapy.
* Any major surgical procedure or radiation within 4 weeks of first study treatment
* Active liver disease, including viral or other hepatitis, or cirrhosis
* Pregnancy or lactation
* Active hepatitis or other active infections
* Any other significant medical condition not under control, including any acute coronary syndrome within the past 6 months.
* Patients with a permanent pacemaker
* Patients with a QTcF or QTcB > 480 ms in the baseline EKG
* Systemic corticosteroids (e.g. prednisone ≥ 12.5 mg/day or dexamethasone ≥ 2 mg/day) for the purpose of palliating tumor-related symptoms will not be allowed within 1 week of starting treatment on trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-07-06 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
To assess the safety of PU-H71 in patients with advanced malignancies. | 2 years
  Toxicity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.0. All patients enrolled who receive study drug will be eligible for these analyses.
To assess the tolerability of PU-H71 in patients with advanced malignancies. | 2 years
  Toxicity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.0.
To assess the pharmacokinetics of PU-H71 in patients with advanced malignancies. | The investigators anticipate these time points to be: 5 min (+mins), 3-4, 18-24 and 44-48 hours post-injection.
  Blood will be drawn at the multiple time points for radioactive pharmacokinetic and metabolite analyses of 124I-PUH71
To determine the maximum tolerated dose (MTD) based on toxicity analysis. | 2 years
  Toxicity will be monitored using NCI- Common Terminology Criteria for Adverse Events version (4.0).Patients receiving at least 3 out of 4 planned doses of study drug developing a drug-related toxicity will be eligible for these analyses.

SECONDARY OUTCOMES:
To assess anti-tumor activity as defined by response rate | 2 years
  complete response (CR), partial response (PR), stable disease (SD), duration of response, and progression free survival (PFS). Patients with measurable disease will be eligible for these analyses.
To evaluate 124I-PU-H71 as a non-invasive means to determine tumor pharmacokinetics and intra-tumoral concentration | 2 years
  In a selected group of patients with advanced malignancies. All patients who undergo planned imaging will be eligible for this analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Komal Jhaveri, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm